# **Statistical Analysis Plan**

NCT04448847

**Document date: 12-FEB-2021** 

Chr. Hansen A/S Trial Id: HND-GI-036 Author: AH

Statistical Analysis Plan

Date: Version No.:

Status:

Page:

4. February 2021

v1.0 FINAL




# Statistical Analysis Plan

# Title:

Discovering the mechanisms of action for the in-vivo protection of Aspirin-induced enteropathy by Bifidobacterium breve Bif195 in man - a randomized, double-blinded, placebo-controlled, cross-over trial in healthy volunteers

Trial Id: HND-GI-036

Author: AH

Statistical Analysis Plan

Date: Version No.: 4. February 2021

Version No.: Status:

Page:

FINAL




# Trial participants:

Principal Investigator:

Filip Krag Knop

Center for Klinisk Metabolisk forskning, Gentofte Hospital

Sponsor's representative

Anders Damholt

Head of Clinical Development, Human Health Innovation,

Chr. Hansen A/S

Trial Statistician:

Andreas Habicht

Senior Statistician, Signifikans Aps

Author: AH Statistical Analysis Plan Date:

Version No.:

4. February 2021

Status: Page: FINAL 3 of 15




# Signature page:

| Sponsor's representative: | | |
|--------------------------------|-----------------|-----------------------|
| Docusigned by: Anders Damkolt | Anders Damholt | 12-Feb-21 13:52 CET |
| Signature: | Print Name: | Date: |
| Principal Investigator: | | |
| Pilip trag tuop | Filip Krag Knop | 12-feb-21 10:00 EST |
| Signature: | Print Name: | Date: |
| Trial Statistician: | | |
| Docusigned by: Andras Habicut | Andreas Habicht | 12-Feb-21 13:29 CE |
| Signature: | Print Name: | Date: |

Chr. Hansen A/S Trial Id: HND-GI-036 Author: AH

Statistical Analysis Plan

Date: Version No.: Status: Page:

4. February 2021 FINAL




# Content

| Cor | itent | | 4 |
|---|---|---|---|
| List | of Abbrev | riations | 5 |
| 1 | Introdu | ction and Summary | 7 |
| | 1.1 | Introduction | 7 |
| | 1.2 | Summary | 7 |
| | Prima | ary and Secondary Outcome Variables | 8 |
| 2 | Trial O | Trial Objective | |
| | 2.1 | Primary Objectives | 9 |
| | 2.2 | Secondary Objectives | 9 |
| 3 | 3 Trial Design | | |
| 4 | Trial Population | | |
| 5 | Statistical Methodology | | |
| | 5.1 | 5.1 General statistical considerations | |
| | 5.2 | Subject disposition | 11 |
| | 5.3 | Handling of Missing Data and Dropouts | 12 |
| | 5.4 | Primary Efficacy Outcome Variable | |
| | 5.5 | Secondary Safety Outcome Variables | |
| | 5.6 | Secondary Efficacy Outcome Variables | 13 |
| | 5.7 | Sensitivity analysis on secondary variables | 13 |
| | 5.8 | Data structure prior primary and secondary analysis | 13 |
| | 5.9 | Challenge analysis | 14 |
| | 5.10 | Other Efficacy Outcome Variable | 15 |
| | 5.11 | Control of Multiplicity for the Primary and secondary Efficacy Analysis | |
| | 5.12 | Subject Disposition, Demographics and Other Characteristics | 15 |
| 6 | | re | |
| 7 | Refere | nces | 15 |

Author: AH

Statistical Analysis Plan

Date: Version No.:

Status:

Page:

4. February 2021

v1.0

FINAL 5 of 15




#### List of Abbreviations

| AE | Adverse Event |
|-----|-----------------------|
| AOM | Acute Otitis Media |
| AUC | Areas under the curve |
| BMI | Body mass index |
| CFU | Colony Forming Units |

CI Confidence Interval
CRA Clinical Research Associate

CRO Contract Research Organization

CV Coefficient of Variation

eCRF Electronic Case Report Form

EFSA European Food Safety Authority

ePRO Electronic Patient Reported Outcome

FAO Food and Agricultural Organization

FAS Full- analysis set

FDA US Food and Drug Administration

GCP Good Clinical Practice

GDPR General Data Protection Regulation

GI Gastrointestinal
GP General Practitioner

GRAS Generally Regarded as Safe Guardian Parent or Legal Guardian

HR Hearth rate

ICH International Conference on Harmonisation

IEC Independent Ethics Committee
IRB Institutional Review Board

Mg Milligram

LRTI Lower Respiratory Tract Infections

Min Minutes
mL Milliliter
N Sample Size

PI Principle Investigator

PP Per protocol
QC Quality Control

Author: AH

Statistical Analysis Plan

Date:

4. February 2021

Version No.:

FINAL

Status: Page:


Sıgnıfıkans

QPS Qualified Presumption of Safety

QQ Quantiles-Quantiles RA Regulatory Authority

RTI Respiratory Tract Infections

SAE Serious Adverse Event
SAP Statistical Analysis Plan
SAS Safety Analysis Set
SD Standard Deviation

URTI Upper Respiratory Tract Infections

WHO World Health Organization

Date: Version No.: Status: Page: 4. February 2021 v1.0 FINAL 7 of 15




# 1 Introduction and Summary

#### 1.1 Introduction

The present Statistical Analysis Plan (SAP) describes in detail and in accordance with ICH-GCP guidelines (1) and Signifikans Aps SOPs the statistical analyses to be carried out for the HND-GI-036 trial.

# 1.2 Summary

The table below provide an overview of all analyses performed on the primary, secondary and exploratory endpoints.

Author: AH Statistical Analysis Plan Date:

4. February 2021

v1.0

Status: Page:

Version No.:

FINAL




# Primary and Secondary Outcome Variables

| Variables | Time point | Endpoint | Analysis performed |
|---|---|---|---|
| Primary Week 2, 3 4 and 5 Lanza score | | Lanza score | Generalized Estimating |
| outcome | | | Equations (GEE) model |
| variables | | | including the following |
| | | | terms: Treatment (Bif195 |
| | | | or Placebo), Sequence |
| | | | (First Bif195 or Placebo), |
| | | | Period (1 and 2) and |
| | | | baseline (visit 2) value |
| Secondary | Week 2, 3 4 and 5 | Blood safety | Each parameter will be |
| outcome | 1000 | parameters: | analysed using a proc |
| variables | | Creatinin, Potasium, | mixed model with patient |
| (safety and | | Sodium, ALAT, ASAT, | as Random effect. The |
| efficacy) | | HbA1c, Glucose (from | following terms will be |
| | | HbA1c), CRP, | including in the model: |
| | | Leucocytes, | Treatment (Bif195 or |
| | | Thrombocytes | Placebo), Sequence (First |
| | | Blood efficacy | Bif195 or Placebo), Period |
| | | parameters: | (1 and 2) and baseline |
| | | Erytrocytes, | (visit 2) value |
| | | Haematocrit, | |
| | | Haemoglobin, INR | |

Author: AH Statistical Analysis Plan Version No.:

Status:

Page:

4. February 2021

VI.0 FINAL




# 2 Trial Objective

## 2.1 Primary Objectives

Clinical evaluation of stomach and duodenum via the (5-scale) Lanza score.

0 = no visible lesions

1 = redness and hyperemia in mucosa

2 = 1 or 2 erosions or hemorrhaging lesions

3 = 3-10 erosions of hemorrhaging lesions

4 = >10 erosions or hemorrhaging lesions or

an ulcer

Erosions = mucosal disruption denuded of villi with or w/o exudates or red color Ulcer = large erosion with central area with exudates Ref: Soylu et al. 2008, World J Gastroenterol, 14(43), 6704-6710

#### 2.2 Secondary Objectives

Safety blood parameters:

Blood safety parameters: Creatinin, Potasium, Sodium, ALAT, ASAT, HbA1c, Glucose (from HbA1c), CRP, Leucocytes, Thrombocytes

Efficacy blood parameters:

Erytrocytes, Haematocrit, Haemoglobin, INR

Author: AH Statistical Analysis Plan Date:

4. February 2021

v1.0

Status: Page:

Version No.:

FINAL 10 of 15




# 3 Trial Design

# Study design (HND-GI-036)

- Aspirin 300 mg/day (1 capsule at breakfast)
- Placebo or 100 B CFU Bif195/day (1 capsule at breakfast, 1 capsule in the evening)



Chr. Hansen A/S Trial Id: HND-GI-036 Author: AH

Statistical Analysis Plan

Date: Version No.:

Status:

Page:

4. February 2021 v1.0

1




# 4 Trial Population

For the statistical analysis, the randomized subjects will be divided into the following datasets:

Full Analysis Set (FAS):

Subjects who are randomized and have consumed at least one dose of study product and for whom efficacy data is available.

No response to challenge
Subjects not responding on the Aspirin challenge response defined as having Lanza score=0 on all visits (visits 2, 3 4 and 5)

Modified FAS (mFAS)

FAS population minus NC population.

Per Protocol Set (PPS)

Subjects, who are randomized and have consumed at least one dose of study product, have available efficacy data and have no major protocol deviations

All endpoints will be analyzed on the FAS populations. For sensitivity analysis, selected analyses will also be performed on the mFAS and PPS.

# 5 Statistical Methodology

#### 5.1 General statistical considerations

All statistical tests will be assessed using a nominal two-sided significance level of 5%.

The two treatment groups will be labelled as Bif195 and Placebo.

Weeks will be calculated as number of days divided by 7 Months will be calculated as number of days divided by 30.4375 Years will be calculated as number of days divided by 365.25

Number of days will be calculated using end date minus start date +1.

#### 5.2 Subject disposition

An overall summary table of the subject disposition will be prepared with number of patients in the following categories (and sub-categories):

- Screened and randomized patients
- Analysis populations (FAS and mFAS)
- End of study reason

Version No.: Status: Page: 4. February 2021 v1.0 FINAL 12 of 15

Sıgnıfıkans


## 5.3 Handling of Missing Data and Dropouts

No imputation of data will be carried out in case of missing data, but all available data will be used.

#### 5.4 Primary Efficacy Outcome Variable

Primary efficacy variable: Lanza score ranging from 0 (no visible lesions) to 4.

Change form baseline prior each period will be calculated and used in the analysis i.e. (visit 3 minus visit 2) (visit 5 minus visit 4).

This ordinal endpoint will be analysed using a Generalized Estimating Equations (GEE) model including the following terms:

- Treatment (Bif195 or Placebo)
- Sequence (first Bif195 or Placebo)
- Period (1 and 2)
- Baseline (visit 2) value

The model will take in to account the crossover design of the study with same patients having a result after both treatments.

- 1) Firstly, the analyse will include terms of Treatment, Sequence, period and baseline (visit 2) value
- If no significant terms of either sequence or period, the factors will be removed from the model prior evaluating treatment effect

#### 5.5 Secondary Safety Outcome Variables

Secondary safety outcome variables: Blood safety parameters: Creatinin, Potasium, Sodium, ALAT, ASAT, HbA1c, Glucose (from HbA1c), CRP, Leucocytes, Thrombocytes

Each parameter will be analysed using a proc mixed model with patient as Random effect.

Sequence and period effect will be evaluated prior evaluating the treatment effect in a similar way as the primary efficacy outcome variable.

For statistical analysis of data measured on an interval scale model check is assessed using QQ residual plots together with Kolmogorov-Smirnov test for normality.

In case for normality not reached using untransformed data nor transformed data using the log2-scale, appropriate non-parametric statistical methods will be used instead.

 Date:
 4. February 2021

 Version No.:
 v1.0

 Status:
 FINAL

 Page:




# 5.6 Secondary Efficacy Outcome Variables

Secondary Efficacy outcome variables: Erytrocytes, Haematocrit, Haemoglobin, INR. All variables are analysed like the secondary safety outcome variable analysis.

## 5.7 Sensitivity analysis on secondary variables

Percent change from baseline on the above secondary variables will also be analysed, where baseline value prior each period (visit 2 and visit 4) is set to index=100.

Subject 1, visit 2 = 1.2 (index=100)

Subject 1, visit 3 = 3.4 (index=283.3, calculated as 100\*3.4/1.2)

Subject 1, visit 4 = 2.3 (index=100)

Subject 1, visit 5 = 1.0 (index=43.5, calculated as 100\*1.0/2.3)

# 5.8 Data structure prior primary and secondary analysis

Below is the required data structure for using the statistical models (A and B are the two treatment groups).

| subject | sequence | period | tmt | result | baseline |
|---------|----------|--------|-----|--------|----------|
| | 1 AB | 1 | A | 3 | 0 |
| | 1 AB | 2 | В | 5 | 1 |
| 2 | 2 AB | 1 | В | 4 | 4 |
| 2 | 2 AB | 2 | Α | 5 | 3 |
| | 3 AB | 1 | В | 4 | 0 |
| | 3 AB | 2 | A | 3 | 0 |
| 4 | 4 AB | 1 | В | 0 | 2 |
| 4 | 4 AB | 2 | A | 3 | 0 |
| | 5 AB | 1 | Α | 4 | 0 |
| | 5 AB | 2 | В | 1 | 0 |
| ( | 5 BA | 1 | A | 3 | 0 |
| 6 | 5 BA | 2 | В | 4 | 1 |
| 7 | 7 BA | 1 | В | 3 | 0 |
| | 7 BA | 2 | A | 2 | 0 |
| 8 | B BA | 1 | В | 4 | 0 |
| 8 | B BA | 2 | A | 4 | 0 |
| 9 | BA | 1 | Α | 1 | 1 |
| 9 | 9 BA | 2 | В | 2 | 0 |
| 10 | BA | 1 | Α | 2 | 1 |
| 10 | BA | 2 | В | 4 | 2 |

Chr. Hansen A/S
Trial Id: HND-GI-036
Author: AH
Statistical Analysis Plan

Date: 4. February 2021
Version No.: v1.0
Status: FINAL
Page: 14 of 15


# 5.9 Challenge analysis

The challenge model will be analysed comparing baseline (visit 2 and 4) with "after" results (visit 3 and visit 5) using similar model as the primary and secondary outcome analysis with the following terms in the model:

- Treatment (Bif195 or Placebo)
- Sequence (first Bif195 or Placebo)
- Period (1 and 2)
- Before\_after (baseline and "after")

The challenge model will thereby be analysed adjusted for period, sequence and treatment.

The data will be structured as seen below:

| subject | sequence | period | tmt | Before_after | result |
|---------|----------|--------|-----|--------------|--------|
| 1 | AB | 1 | Α | before | 1 |
| 1 | AB | 1 | Α | after | 2 |
| 1 | AB | 2 | В | before | 1 |
| 1 | AB | 2 | В | after | 0 |
| 2 | 2 AB | 1 | В | before | 4 |
| 2 | 2 AB | 1 | В | after | 5 |
| 2 | 2 AB | 2 | Α | before | 4 |
| 2 | 2 AB | 2 | Α | after | 5 |
| 3 | B AB | 1 | В | before | 4 |
| 3 | B AB | 1 | В | after | 3 |
| 3 | B AB | 2 | Α | before | 4 |
| 3 | B AB | 2 | Α | after | 3 |
| 4 | AB | 1 | В | before | 0 |
| 4 | 4 AB | 1 | В | after | 3 |
| 4 | 4 AB | 2 | Α | before | 0 |
| 4 | 4 AB | 2 | A | after | 3 |
| Ę | AB | 1 | Α | before | 4 |
| Ę | AB | 1 | Α | after | 1 |
| | 5 AB | 2 | В | before | 4 |
| Ę | 5 AB | 2 | В | after | 1 |
| • | S BA | 1 | Α | before | 3 |
| • | BA BA | 1 | Α | after | 4 |
| • | 6 BA | 2 | В | before | 3 |
| 6 | BA | 2 | В | after | 4 |
| 7 | 7 BA | 1 | В | before | 3 |
| 7 | 7 BA | 1 | В | after | 2 |
| 7 | 7 BA | 2 | Α | before | 3 |
| 7 | 7 BA | 2 | A | after | 2 |

Date: Version No.: Status: 4. February 2021 v1.0 FINAL 15 of 15




## 5.10 Other Efficacy Outcome Variable

All biopsies will be collected and analysed post unblinding of the study. Data will be analysed descriptively.

## 5.11 Control of Multiplicity for the Primary and secondary Efficacy Analysis

No adjustment for multiplicity is done.

# 5.12 Subject Disposition, Demographics and Other Characteristics

Subject disposition demographics and other characteristics will be reported descriptively.

## 6 Software

All statistical analyses will be computed using the statistical software SAS®, Release 9.3 or later versions.

## 7 References

- Slides set: 2021-01-12 Strain X MoA study.pptx
- Bif195 study group meeting\_29Jan2020\_NL\_genskabt.pptx

